CLINICAL TRIAL: NCT04505904
Title: A Pull to be Close: the Differentiating Effects of Oxytocin and Grief Stimulus Type on Approach Behavior in Complicated Grief
Brief Title: Oxytocin and Approach-avoid in Grief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Basic Science
Other Study IDs: CGOT1620
Record Dates: First submitted 2020-08-04; First posted 2020-08-10 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Prolonged Grief Disorder; Bereavement
Keywords: Oxytocin; Approach/Avoid; Older adults; Complicated Grief
MeSH Terms: conditions — Prolonged Grief Disorder | interventions — Oxytocin

ARMS (2):
- Syntocinon First (Experimental): Crossover design, all participants received experimental condition at either visit one or visit two, and the placebo at the other visit. This arm designates those who received syntocinon at visit one and placebo at visit two. Syntocinon is 24 IU dose administered intranasally in spray form.
  Interventions: Drug: Syntocinon; Drug: Placebo
- Placebo First (Placebo Comparator): Crossover design, all participants received experimental condition at either visit one or visit two, and the placebo at the other visit. This arm designates those who received placebo at visit one, and syntocinon at visit two.
  Interventions: Drug: Syntocinon; Drug: Placebo

INTERVENTIONS:
Drug: Syntocinon — Synthetic oxytocin spray, 24 IU per spray.
Drug: Placebo — Placebo spray with no active ingredient.

SUMMARY:
This is a completed project which was initiated prior to January 18,2017

Background: Theoretical models of complicated grief (CG) suggest that maladaptive approach (e.g., perseverative proximity-seeking of the deceased) or avoidance (e.g., excessive avoidance of reminders) behaviors interfere with a person's ability to integrate the loss and recover from their loved one's death. Due in part to conflicting evidence, little mechanistic understanding of how these behaviors develop in grief exists. We sought to (1) identify behavioral differences between CG and non-CG groups based on implicit bias for grief-, deceased-, and social-related stimuli, and (2) test the role of the neuropeptide oxytocin in shaping approach/avoidance bias.

Methods: Widowed older adults with and without CG completed an approach/avoidance task measuring implicit bias for personalized, non-specific, grief-related, and other stimuli. In a double-blinded, randomized, counterbalanced design, each participant attended both an intranasal oxytocin session and a placebo session. Aims were to (1) identify differential effects of CG and stimulus type on implicit approach/avoidance bias [placebo session], and (2) investigate interactive effects of CG, stimulus type, and oxytocin vs. placebo on approach/avoidance bias [both sessions].

ELIGIBILITY:
Inclusion Criteria:

• Adult individual experiencing death of a spouse or partner between 6 and 36 months prior to enrollment

Exclusion Criteria:

* Inability to comprehend English;
* medical contraindications for other components of the study,
* active suicidality
* active homicidality
* active psychotic symptoms
* ongoing major health conditions such as cancer; uncontrolled hypertension; and medications likely to impact the oxytocin system (e.g., systemic corticosteroids).
* pregnant status or suspected pregnant status
* premenopausal status

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- With Complicated Grief: Syntocinon First, Then Placebo: Crossover design. This arm designates the Complicated grief group, as designated to >=25 cutoff score on standardized measure (the Inventory of Complicated Grief) who received experimental condition at visit one, and placebo at visit two 7-10 days later.
  Syntocinon: Synthetic oxytocin spray, 24 IU per spray.
  Placebo: Placebo spray with no active ingredient.
- With Complicated Grief: Placebo First, Then Syntocinon: Crossover design. This arm designates the Complicated grief group, as designated to >=25 cutoff score on standardized measure (the Inventory of Complicated Grief) who received placebo condition at visit one, and syntocinon at visit two 7-10 days later.
  Syntocinon: Synthetic oxytocin spray, 24 IU per spray.
  Placebo: Placebo spray with no active ingredient.
- Without Complicated Grief: Syntocinon First, Then Placebo: Crossover design. This arm designates the Non-Complicated grief group, as designated to <25 cutoff score on standardized measure (the Inventory of Complicated Grief) who received experimental condition at visit one, and placebo at visit two 7-10 days later.
  Syntocinon: Synthetic oxytocin spray, 24 IU per spray.
  Placebo: Placebo spray with no active ingredient.
- Without Complicated Grief: Placebo First, Then Syntocinon: Crossover design. This arm designates the Non-Complicated grief group, as designated to <25 cutoff score on standardized measure (the Inventory of Complicated Grief) who received placebo condition at visit one, and experimental condition at visit two 7-10 days later.
  Syntocinon: Synthetic oxytocin spray, 24 IU per spray.
  Placebo: Placebo spray with no active ingredient.
Period: Overall Study
Arm/Group | With Complicated Grief: Syntocinon First, Then Placebo | With Complicated Grief: Placebo First, Then Syntocinon | Without Complicated Grief: Syntocinon First, Then Placebo | Without Complicated Grief: Placebo First, Then Syntocinon
Started | 11 | 11 | 11 | 11
Completed | 9 | 8 | 11 | 11
Not Completed | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Complicated Grief: Crossover design, all participants received experimental condition at either visit one or visit two, and the placebo at the other visit. This arm designates the Complicated grief group, as designated to >25 cutoff score on standardized measure (the Inventory of Complicated Grief). All participants in this group received both synthetic oxytocin and placebo
  Syntocinon: Synthetic oxytocin spray, 24 IU per spray.
  Placebo: Placebo spray with no active ingredient.
- Noncomplicated Grief: Crossover design, all participants received experimental condition at either visit one or visit two, and the placebo at the other visit. This arm designates the noncomplicated grief group, as divided based on cutoff score on standardized measure (the Inventory of Complicated Grief)
  Syntocinon: Synthetic oxytocin spray, 24 IU per spray.
  Placebo: Placebo spray with no active ingredient.
- Total: Total of all reporting groups
Arm/Group | Complicated Grief | Noncomplicated Grief | Total
Number analyzed (Participants) | 17 | 22 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.96 (6.68) | 69.83 (6.68) | 69.45 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 19 | 28
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 15 | 22 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 22 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 22 | 39
Inventory of Complicated Grief [Mean (Standard Deviation); unit: units on a scale] — Total score range: 0-76, with higher score meaning higher symptom severity/burden.
  units on a scale | 35.18 (7.9) | 14.47 (6.36) | 23.5 (7.0)
Beck Depression Inventory - II [Mean (Standard Deviation); unit: units on a scale] — Range is 0 (absent) to 30 (highest possible symptom score, highest depression severity). Total Score is reported here.
  units on a scale | 16.41 (6.7) | 6 (4.86) | 10.4 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time (ms) of a Push or Pull of a Joystick in a Standard Interactive Approach/Avoid Task.
Description: Participants completed the approach avoid task twice per session, with reversed instructions on the second run (i.e., "pull for yellow" became "push for yellow"). Each seven-minute run of the task consisted of 144 2500ms trials (288 trials per visit, 576 trials total across runs/sessions; 500ms inter-trial-interval). Order of instructions (i.e., "push yellow" vs. "pull yellow") was randomized and counterbalanced across participants and sessions, to address potential for order effects/habituation. Stimuli were presented via Inquisit 4 (2014), in a pseudorandomized order determined by genetic algorithm (Wager & Nichols, 2003).
  Relative approach/avoidance bias was computed by subtracting median response time (RT; latency to joystick full extension) on PULL/approach trials in each stimulus category from PUSH/avoid trials in the same category (Rinck & Becker, 2007). Positive response bias values indicate relative approach bias; negative values indicate relative avoidance bias.
Time Frame: 120 minutes
Population: Of note, for analysis purposes, we collapsed across crossover groups to yield two groups, complicated grief and non-complicated grief. This is consistent with reporting methods of other relevant literature in this area and allows for direct conceptual comparison to these previous studies.
Measure: Mean (Standard Deviation); unit: Milliseconds (contrast score)
Groups:
- With Complicated Grief: Those with > =25 score on ICG
- Noncomplicated Grief Group: Those scoring < 25 score on Inventory of Complicated Grief (ICG).
Arm/Group | With Complicated Grief | Noncomplicated Grief Group
Number analyzed (Participants) | 17 | 22
Milliseconds (contrast score)
  Syntocinon First: number analyzed (Participants) | 9 | 11
  Syntocinon First | 29 (21) | 18 (18.9)
  Placebo First: number analyzed (Participants) | 8 | 11
  Placebo First | 7.5 (21) | 13.0 (11.5)

ADVERSE EVENTS:
Time Frame: 6 hours per participant (two visits of three hours each). Participants were monitored for any adverse even to nasal spray during laboratory visit for data collection.
Description: All adverse events encountered in this study are classified as "other" as they are not serious or all-cause mortality.
Groups:
- Syntocinon: Participants with adverse event during syntocinon condition
- Placebo: Participants with adverse events during placebo condition
Arm/Group | Syntocinon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 2/39 | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Syntocinon (N=39) | Placebo (N=39)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant discontinued functional MRI data collection due to nausea while in the scanner.
Back pain (General disorders) | 0 (0) | 1 (1) — Participant experienced back pain while in the MRI scanner. Participant chose to discontinue study participation due to back pain.
Incidental Finding (General disorders) | 1 (1) | 0 (0) — There was an incidental radiologic finding requiring follow-up by participant's primary care physician. Participant discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT04505904/Prot_SAP_001.pdf